CLINICAL TRIAL: NCT07238387
Title: Evaluation of Nystagmus Examinations Conducted Using Wearable Augmented Reality Glasses in Vertigo Patients: A Randomized Equivalence Study
Brief Title: Evaluation of Nystagmus Examination Using Wearable AR Glasses in Vertigo Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 202500606B0
Record Dates: First submitted 2025-09-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Vertigo; Vestibular Disorder; Nystagmus
MeSH Terms: conditions — Vertigo; Vestibular Diseases; Nystagmus, Pathologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR-First Examination Sequence (Experimental): AR-based examination first, then conventional examination
  Interventions: Device: Wearable Augmented Reality Glasses for Nystagmus Examination; Device: Conventional Nystagmus Examination
- Conventional-First Examination Sequence (Active Comparator): Conventional examination first, then AR-based examination
  Interventions: Device: Wearable Augmented Reality Glasses for Nystagmus Examination; Device: Conventional Nystagmus Examination

INTERVENTIONS:
Device: Wearable Augmented Reality Glasses for Nystagmus Examination — Intervention 1 - Wearable Augmented Reality Glasses for Nystagmus Examination Participants undergo a standardized nystagmus examination using wearable augmented reality (AR) glasses equipped with an integrated eye-tracking system. The AR-based system records real-time eye movements in both light and dark conditions, allowing for simultaneous examiner visualization and data storage. This method eliminates the need for traditional Frenzel goggles and provides automated signal quality assessment.
Device: Conventional Nystagmus Examination — Intervention 2 - Conventional Nystagmus Examination Participants undergo a conventional clinical nystagmus examination performed by an otolaryngologist using standard Frenzel goggles under similar test conditions. Eye movements are visually assessed without integrated digital recording or automated signal analysis.

SUMMARY:
Background and Purpose:

Vertigo is common in emergency and outpatient settings, yet standard oculomotor testing usually requires dedicated equipment and exam rooms. This study evaluates whether nystagmus examinations performed with wearable augmented-reality (AR) glasses are equivalent to conventional examination-room testing for classifying central vs. peripheral vertigo. The investigators also assess diagnostic accuracy, patient tolerability, and the reliability of AR-based interpretation (test-retest and inter-rater).

Study Design:

Prospective, single-center, within-subject randomized equivalence study at Kaohsiung Chang Gung Memorial Hospital. Each participant completes both AR-based and conventional oculomotor testing in a randomized order during the same visit, separated by a 30-minute washout. The study uses an evaluator-blind approach: de-identified trajectories are reviewed offline by independent experts who are masked to test modality. A follow-up visit (~1 week) captures adverse events and patient experience.

Participants:

Adults (≥18 years) presenting with vertigo who can tolerate the AR headset and provide consent. Key exclusions include conditions that prevent reliable eye-tracking (e.g., corrected visual acuity <20/40), recent use of vestibular suppressants (within 24 hours), and other factors limiting cooperation or safety.

Interventions and Procedures:

The AR system records eye movements and presents standardized visual stimuli. Conventional testing follows current clinical standards (e.g., Frenzel/oculomotor exam). All recordings are stored securely for blinded review.

Outcomes:

Primary endpoint: Equivalence of diagnostic agreement (central vs. peripheral) between AR-based and conventional methods, quantified by Cohen's kappa (κ) with a predefined equivalence margin.

Secondary endpoints: (1) Diagnostic accuracy of the AR method in a clinically-indicated imaging subgroup (MRI preferred; CT as needed) using a sequential evaluation strategy; (2) Patient discomfort/tolerability using VAS and CSQ-VR, compared between modalities; (3) Test-retest reliability of AR-based classifications; (4) Inter-rater reliability between independent evaluators, with a third reader adjudicating discordant cases; (5) prespecified subgroup analyses by age, medical history, and vestibular function.

Sample Size and Duration:

Approximately 200 participants will be enrolled (target ~180 evaluable after ~10% attrition). Total study duration is ~2 years, including enrollment, follow-up, and analysis.

Risks and Benefits:

Both tests are non-invasive. Potential transient discomfort (e.g., eye strain or cybersickness) will be monitored. There may be no direct benefit to participants; however, results could support broader, more accessible, and standardized vertigo assessment.

Data Security and Privacy:

All data are de-identified, stored on secure platforms with role-based access and audit trails. Safety events are monitored and graded, and protocol deviations are handled per Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with vertigo/dizziness suggestive of a central or peripheral vestibular disorder.
* Able to complete both AR-based and conventional oculomotor testing during the same visit (with ~30-minute washout).
* Provide written informed consent.
* Adequate vision for eye-tracking and calibration (e.g., corrected visual acuity ≥20/40 in each eye).
* Willing and able to return for the follow-up visit.

Exclusion Criteria:

* Use of vestibular-suppressant medications within 24 hours prior to testing (e.g., benzodiazepines, antihistamines, anticholinergics).
* Ocular conditions that would interfere with reliable eye tracking (e.g., corrected visual acuity <20/40, dense cataract, severe ptosis/strabismus, active ocular infection/inflammation).
* History of photosensitive epilepsy or seizure disorder triggered by visual stimuli.
* Severe motion sickness/cybersickness or inability to tolerate the AR headset.
* Significant cognitive impairment or psychiatric condition precluding informed consent or protocol compliance.
* Pregnant or breastfeeding (per investigator judgment and IRB policy).
* Any other condition that, in the investigator's opinion, would make participation unsafe or confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Equivalence of Diagnostic Agreement (Central vs Peripheral) Between AR-Based and Conventional Examinations, Assessed by Cohen's Kappa | Day 1 (immediately after completion of both AR-based and conventional examinations)
  Cohen's Kappa (κ) will be used to evaluate diagnostic agreement between AR-based and conventional examinations. κ ranges from -1.0 to 1.0, where 1.0 indicates perfect agreement, 0 indicates chance-level agreement, and negative values indicate worse-than-chance agreement. Higher κ values represent better diagnostic consistency.

SECONDARY OUTCOMES:
Diagnostic Accuracy of AR-Based Examination Compared to Neuroimaging (Sensitivity, Specificity, PPV, NPV) | Within 30 days after Day 1 (baseline examination), for participants undergoing clinically indicated MRI (preferred) or CT
Test-Retest Reliability of AR-Based Examination (Cohen's Kappa) | Day 1 - within 1 hour after completion of the initial AR-based examination
  Test-retest reliability of AR-based examination will be assessed using Cohen's Kappa coefficient (κ). κ ranges from -1.0 to 1.0, where 1.0 indicates perfect agreement, 0 indicates chance-level agreement, and negative values indicate worse-than-chance agreement. Higher κ values indicate better reliability.
Patient Discomfort Measured by Visual Analog Scale (VAS) | Day 1 - immediately after completion of AR-based and conventional examinations
  Visual Analog Scale (VAS) will be used to assess patient-reported discomfort immediately after each test. The VAS ranges from 0 to 10, where 0 indicates no discomfort and 10 indicates the worst imaginable discomfort. Higher scores represent greater discomfort.
Patient Discomfort Measured by Cybersickness Questionnaire for Virtual Reality (CSQ-VR) | Day 1 - immediately after completion of AR-based and conventional examinations
  Patient discomfort will also be measured using the Cybersickness Questionnaire for Virtual Reality (CSQ-VR). The CSQ-VR assesses cybersickness symptoms across multiple domains (e.g., nausea, oculomotor strain, disorientation). Scores range from 6 to 42, with higher scores indicating more severe discomfort.
Inter-Rater Reliability of Diagnostic Interpretations (Cohen's Kappa; Fleiss' Kappa if applicable) | Following Day 1 (baseline visit), blinded offline review of examination recordings prior to database lock
  Inter-rater reliability of diagnostic interpretations will be assessed using Cohen's Kappa coefficient (κ) for two raters, and Fleiss' Kappa for three or more raters.
  Cohen's Kappa (κ): Ranges from -1.0 to 1.0, where 1.0 indicates perfect agreement, 0 indicates agreement equivalent to chance, and negative values indicate worse-than-chance agreement. Higher values represent better inter-rater reliability.
  Fleiss' Kappa: Ranges from -1.0 to 1.0, with the same interpretation as Cohen's Kappa.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results will be made available to qualified researchers upon reasonable request. Data will be shared beginning 6 months after publication of the main results and for up to 5 years thereafter. Requests should be directed to the principal investigator via institutional email and must include a methodologically sound proposal and a signed data use agreement.